CLINICAL TRIAL: NCT07307989
Title: Early Statin-Ezetimibe Combination vs. Statin Monotherapy to Achieve LDL-C < 70 mg/dL in Recent Ischemic Stroke Patients With Evidence of Atherosclerosis: A Randomized Controlled Trial
Brief Title: Early Statin-Ezetimibe Combination vs. Statin Monotherapy in Stroke With Atherosclerosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Chang Gung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NSTC 114-2314-B-182-019-
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Ischemic Stroke; Hypercholesteremia
Keywords: ischemic stroke; hypercholesteremia; statin; ezetimibe
MeSH Terms: conditions — Ischemic Stroke; Hypercholesterolemia | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Ezetimibe; Rosuvastatin Calcium; Atorvastatin

STUDY DESIGN:
Intervention Model Description: To test statin plus ezetimibe vs statin monotherapy to lower LDL-C < 70 mg/dl
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Statin plus ezetimibe (Experimental): Moderate-intensity statin plus ezetimibe as the interventional group. Both fixed-dose combination of statin/ezetimibe, such as Vytorin (simvastatin 20mg/ezetimibe 10mg), Atozet (atorvastatin 20mg/ezetimibe 10mg), Cretrol (rosuvastatin 10mg/ezetimibe 10mg) and one pill of ezetimibe added to moderate-intensity statins are allowed.
  Interventions: Drug: statin + ezetimibe
- Statin monotherapy (Active Comparator): Moderate- or high-intensity statin monotherapy, including atorvastatin 10-80 mg/d, rosuvastatin 5-20 mg/d, pitavastatin 1-4 mg/d
  Interventions: Drug: Statin monotherapy (rosuvastatin or atorvastatin)

INTERVENTIONS:
Drug: statin + ezetimibe — Moderate-intensity statin plus ezetimibe 10mg
  Arms: Statin plus ezetimibe
Drug: Statin monotherapy (rosuvastatin or atorvastatin) — Moderate- or high-intensity statin monotherapy
  Arms: Statin monotherapy

SUMMARY:
This study will be conducted at six medical institutions in Taiwan, recruiting patients who visit neurology outpatient clinics or are hospitalized within 30 days after an ischemic stroke.

Participants will be randomly assigned to either the experimental group (moderate-intensity statin plus ezetimibe) or the control group (moderate- or high-intensity statin).

Research assistants will screen patients aged 40 or older who have had an ischemic stroke or transient ischemic attack within 30 days, have atherosclerosis, and have LDL-C levels ≥100 mg/dL. Eligible cases will be reviewed by the attending physician. With physician approval, patients will be invited to join the study, and those who agree and sign informed consent will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* (1) clinical diagnosis of ischemic stroke or TIA; (2) Stroke or TIA symptoms and randomized within 30 days, then taking assigned medication within 2 days of randomization; (3) aged 20 years or older; (4) LDL-C ≥ 100 mg/dL after index ischemic stroke or TIA; (5) having evidence of atherosclerosis.

Exclusion Criteria:

* (1) end stage renal disease because there is no clear benefit of LDL-C lowering therapy in these patients; (2) history of statin intolerance; (3) history of ezetimibe intolerance; or (4) ALT > 100 U/L.(5) Statins were regularly used before stroke. (6) Ezetimibe was used before stroke.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
LDL-C levels < 70 mg/dL | 6 months after randomization

SECONDARY OUTCOMES:
LDL-C levels < 70 mg/dL | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Chiayi Branch, Pozi, Taiwan

IPD SHARING:
Plan to Share IPD: No
IRB did not approve sharing data.

REFERENCES:
- [Result] Derynck R, Gelbart WM, Harland RM, Heldin CH, Kern SE, Massague J, Melton DA, Mlodzik M, Padgett RW, Roberts AB, Smith J, Thomsen GH, Vogelstein B, Wang XF. Nomenclature: vertebrate mediators of TGFbeta family signals. Cell. 1996 Oct 18;87(2):173. doi: 10.1016/s0092-8674(00)81335-5. No abstract available. PMID 8861901